CLINICAL TRIAL: NCT04673461
Title: A Multi-country, Randomized, Double-blind, Placebo-controlled Study Investigating the Efficacy and Safety of STA363 at Two Concentrations (60 mg/mL and 120 mg/mL) Compared to Placebo in Patients With Chronic Discogenic Low Back Pain
Brief Title: Study Investigating STA363 Compared to Placebo in Patients With Chronic Discogenic Low Back Pain
Acronym: STA-02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stayble Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STA-02; 2019-004943-54 (EudraCT Number)
Record Dates: First submitted 2020-12-01; First posted 2020-12-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Discogenic Pain
MeSH Terms: interventions — Lactic Acid

STUDY DESIGN:
Intervention Model Description: Three treatment groups:
  * STA363 60 mg/mL
  * STA363 120 mg/mL
  * Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The test and reference IMPs will be identical in appearance. The kits will not contain any other information about treatment. Therefore, all site staff and patients will be blinded at treatment administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STA363 containing 90 mg (60 mg/mL) lactic acid (Experimental): STA363 containing 90 mg (60 mg/mL) lactic acid will be injected into the center of up to two intervertebral discs. Patients with two discs appropriate for treatment will be treated at both affected levels by two separate injections.
  Each patient will have 5 visits to study site and 1 telephone call. The patient's total time in the study will be approximately 61 weeks (~15 months) including an 8-week screening period.
  Interventions: Drug: STA363 containing 90 mg (60 mg/mL) lactic acid
- STA363 containing 180 mg (120 mg/mL) lactic acid (Experimental): STA363 containing 180 mg (120 mg/mL) lactic acid will be injected into the center of up to two intervertebral discs. Patients with two discs appropriate for treatment will be treated at both affected levels by two separate injections.
  Each patient will have 5 visits to study site and 1 telephone call. The patient's total time in the study will be approximately 61 weeks (~15 months) including an 8-week screening period.
  Interventions: Drug: STA363 containing 180 mg (120 mg/mL) lactic acid
- Placebo (Placebo Comparator): Placebo will be injected into the center of up to two intervertebral discs. Patients with two discs appropriate for treatment will be treated at both affected levels by two separate injections.
  Each patient will have 5 visits to study site and 1 telephone call. The patient's total time in the study will be approximately 61 weeks (~15 months) including an 8-week screening period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: STA363 containing 90 mg (60 mg/mL) lactic acid — STA363 (90 mg) will be injected into maximally two pain-generating degenerated intervertebral discs
  Arms: STA363 containing 90 mg (60 mg/mL) lactic acid
Drug: STA363 containing 180 mg (120 mg/mL) lactic acid — STA363 (180 mg) will be injected into maximally two pain-generating degenerated intervertebral discs
  Arms: STA363 containing 180 mg (120 mg/mL) lactic acid
Drug: Placebo — Placebo will be injected into maximally two pain-generating degenerated intervertebral discs
  Arms: Placebo

SUMMARY:
This is a phase IIb, prospective, multi-country, multicenter, randomized, double-blind, placebo-controlled, parallel group study to investigate the efficacy, safety and transformation of NP following single intradiscal injection of STA363 (lactic acid) into one or two IVDs compared to placebo for the treatment of discogenic low back pain. This study will be conducted in Russia, Spain and the Netherlands.

DETAILED DESCRIPTION:
This is a phase IIb, prospective, multi-country, multicenter, randomized, double-blind, placebo-controlled, parallel group study to investigate the efficacy, safety and transformation of NP following single intradiscal injection of STA363 (lactic acid) into one or two IVDs compared to placebo for the treatment of discogenic low back pain. This study will be conducted in Russia, Spain and the Netherlands.

The primary objective is to demonstrate superiority of STA363 over placebo in reducing low back pain as measured by the NRS. A total of 168 patients will be screened in the study with the aim to recruit 126 patients to be randomly allocated to one of the three treatment groups:

Group 1 - 42 patients will receive STA363 containing 90 mg (60 mg/mL) lactic acid Group 2 - 42 patients will receive STA363 containing 180 mg (120 mg/mL) lactic acid Group 3 - 42 patients will receive placebo

The investigational medical product (IMP) will be injected into the center of up to two IVDs. Patients with two discs appropriate for treatment will be treated at both affected levels by two separate injections.

Each patient will have 5 visits to study site and 1 telephone call. The patient's total time in the study will be approximately 61 weeks (~15 months) including an 8-week screening period.

Each patient will perform a screening visit (Visit 1) maximum 60 days before planned treatment. Randomization and treatment will be performed at Visit 2 (Day 1) after confirmation of patient's eligibility for the study. The IMP will be administered, monitored by fluoroscopy or other available method of real-time x-ray imaging to ensure that an injection is correctly placed in the IVD nucleus and that no leakage occurs. Immediately after treatment the patients should remain supine for as long as possible (at least 1 hour). For safety reasons, patients will be allowed to leave the clinic not earlier than 2 hours after the last injection. After leaving the clinic, patients will be offered analgesics and/or other measures according to standard clinical practice. They will also be given advice on restricted physical activity during the first two weeks after injection. Patients should not drive or operate machinery for 12 hours following the treatment procedure.

Patients will be followed up at 1 month (Visit 3/Day 30±7, visit to study site), 3 months (Visit 4/Day 90±7, telephone call), 6 months (Visit 5/Day 180±7, visit to study site) and 12 months (Visit 6/Day 360±7, visit to study site) after treatment. Follow-up MRI will be conducted as part of Visit 5 and Visit 6, to assess the transformation of the NP into connective tissue and other disc characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study related procedures.
2. Male and female patients ≥18 and ≤70 years.
3. Chronic discogenic low back pain present for more than 6 months prior to the screening visit.
4. Insufficient response or lack of response to at least 6 months of non-operative treatment (analgesics and/or anti-inflammatory medications [paracetamol, non-steroidal anti-inflammatory agents (NSAIDs), opioids], physiotherapy, rehabilitation therapy etc.).
5. Patients who meet all the following NRS selection criteria:

   1. Presence of ≥5 pain NRS assessments (entries) for 7 consecutive days.
   2. NRS daily pain scores between 3-9.
   3. Not more than two ratings "3".
6. One or two treatable IVDs of Pfirrmann grade 2 to 3 on MRI at L2/3 to L5/S1 as confirmed by a central reader, AND the following criteria are met:

   1. Treatable IVD(s) must be IVD(s) with the highest Pfirrmann grade observed in the patient (e.g. a patient with one IVD of grade 3 and four IVDs of grade 2 is considered eligible only if IVD of grade 3 will be injected).
   2. Patients with treatable IVD(s) of grade 2 must have all other lumbar discs rated as grade 1.
   3. Not more than two IVDs of grade 3 at any lumbar level.
   4. No IVDs of grade 4 or 5 at any lumbar level.
7. Ability to understand the written and verbal information about the study.

Exclusion Criteria:

1. Treatment with any investigational product within 3 months prior to the screening visit.
2. Patients with more than two painful IVDs.
3. A painful IVD above L2/3 level.
4. Current infection or prior history of spinal infection (e.g., discitis, septic arthritis, epidural abscess) or an active systemic infection.
5. Previous lumbar spine surgery.
6. Previous disc invasive treatment procedures at the affected level(s) (e.g., intradiscal electrothermal therapy, intradiscal radiofrequency thermocoagulation).
7. Evidence of prior lumbar vertebral body fracture or trauma.
8. Need for spinal decompression assessed by the Investigator.
9. Presence of IVD extrusion or sequestration, or other radiologic findings that in the opinion of the investigator disqualify the patient from being included.
10. Spondylolisthesis or retrolisthesis Grade 2 and above or spondylolysis at the index or adjacent level(s).
11. Lumbar spondylitis or other undifferentiated spondyloarthropathy affecting the index IVD.
12. Patients previously included in the study.
13. Patients suffering from psychosomatic pain in the opinion of the Investigator.
14. Leg pain of compressive origin.
15. Patients requiring continuous treatment with warfarin or other anticoagulant therapy.
16. History of significant neurologic or psychiatric disorders including dementia or seizures.
17. Known alcohol and/or drug abuse.
18. Severe intercurrent illness (e.g. rheumatic disease or chronic pain syndrome) or concomitant treatment (e.g. immunosuppressive drugs), which, in the opinion of the Investigator, may put the patient at risk when participating in the study, or affect the patient's ability to take part in the study.
19. Pregnant or lactating females, or intention to become pregnant within the study period.
20. Known allergy to any of the components of the drug product or placebo.
21. Known allergy or intolerance to the contrast agent Omnipaque®.
22. Known opioid allergy or intolerance.
23. Any other condition that, in the opinion of the Investigator, precludes the patient from taking part in this study.
24. Any specific contraindication for MRI such as claustrophobia, intracranial clips or pacemakers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity at 6 months on a Numerical rating scale | 6 months
  Change from baseline at Month 6 in mean pain intensity measured on a Numerical rating scale (minimum value: 0; maximum value: 10) for 7 consecutive days. Lower scores means a better outcome.

SECONDARY OUTCOMES:
Pain intensity at Month 1, Month 3 and Month 12 on a Numerical rating scale | 1 month, 3 months and 12 months
  Change from baseline at Month 1, 3 and 12 in mean pain intensity measured on a Numerical rating scale (minimum value: 0; maximum value: 10) for 7 consecutive days. Lower scores means a better outcome.
Oswestry Disability Index | 1 month, 3 months, 6 months and 12 months
  Change from baseline in Oswestry Disability Index score (minimal-maximal values: 0-100 where a lower number means better outcome) at Month 1, Month 3, Month 6 and Month 12. Lower scores means a better outcome.
EuroQoL 5-dimension 5-level | 1 month, 3 months, 6 months and 12 months
  Change from baseline in EuroQoL 5-dimension 5-level-index at Month 1, Month 3, Month 6 and Month 12. Higher scores means a better outcome.
Nucleus pulposus transformation | 6 and 12 months
  Quantitative changes in nucleus pulposus (NP) water content (reflecting transformation of NP into connective tissue) at Month 6 and Month 12 (T2-weighted magnetic resonance imaging [MRI] and quantification of T2). Lower scores means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Willem Kallewaard, MD, PhD, Principal Investigator — Rijnstate Hospital
Locations (17):
- Netherlands (2):
  - Alrijne Ziekenhuis Leiderdorp, Leiderdorp
  - Rijnstate Hospital Anesthesiology and Pain, Velp
- Russia (11):
  - Belgorod Regional Clinical Hospital of Saint Joasaph, Belgorod
  - Regional Clinical Hospital #3, Chelyabinsk
  - Kirov State Medical University, Kirov
  - Ochapovsky Regional Clinical Hospital #1, Krasnodar
  - Krasnoyarsk Interdistrict Clinical Emergency Hospital, Krasnoyarsk
  - Siberian Research Clinical Center, Krasnoyarsk
  - Privolzhsky Research Medical University, Nizhny Novgorod
  - Bekhterev Psychiatry and Neurology Center, Saint Petersburg
  - LLC MART, Saint Petersburg
  - Smolensk Regional Clinical Hospital, Smolensk
  - Tula Regional Clinical Hospital, Tula
- Spain (4):
  - Hospital Quirónsalud Córdoba, Córdoba
  - Complejo Hospitalario Ruber Juan Bravo, Madrid
  - Hm Puerta Del Sur, Móstoles
  - Hospital Universitario Quirónsalud Madrid, Pozuelo de Alarcón

IPD SHARING:
Plan to Share IPD: No